CLINICAL TRIAL: NCT05454787
Title: Ondexxya for Intravenous Injection 200mg Drug Use Result Investigation (All Case Investigation)
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9603C00001
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Life Threatening Bleeding; Factor Xa Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This survey will be conducted to investigate the status of occurrence of the safety specifications set for "Safety specification" in patients who received Ondexxya Intravenous Injection 200 mg. In addition, this survey will be implemented to understand the followings by collecting safety and effectiveness information under actual use conditions.

DETAILED DESCRIPTION:
This survey will be conducted to investigate the status of occurrence of the safety specifications set for "Safety specification" in patients who received Ondexxya Intravenous Injection 200 mg. In addition, this survey will be implemented to understand the followings by collecting safety and effectiveness information under actual use conditions.

1. Detection of unknown adverse drug reactions
2. Incidence of adverse drug reactions under actual use conditions of the drug
3. Factors that may affect the safety or effectiveness

"Safety specification" Thrombotic events, Infusion reaction, re-bleeding

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with this drug to neutralize the anticoagulant effect of a FXa inhibitor (apixaban, rivaroxaban, or edoxaban) at onset of a life-threatening bleeding episode or a unarrestable bleeding episode.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with this drug to neutralize the anticoagulant effect of a FXa inhibitor (apixaban, rivaroxaban, or edoxaban) at onset of a life-threatening bleeding episode or a unarrestable bleeding episode.
  The patients treated with direct acting Factor Xa inhibitors (apixaban, rivaroxaban or edoxaban tosilate hydrate) to neutralize anticoagulation effect at the time of life threatening bleeding or uncontrolled bleeding during the period of ethical free provision of the drug ( from the date of market authorization to the date of NHI drug price listing ) are also included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions, Incidence of safety specifications, Incidence of adverse drug reactions by patient background factor | 30days
  Incidence of adverse drug reactions, Incidence of safety specifications, Incidence of adverse drug reactions by patient background factor

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — Astrazeneca KK
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli Org.
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/